CLINICAL TRIAL: NCT06947642
Title: Comparison Between Ultrasound-guided Pectoral Nerve Blocks, Thoracic Erector Spinae Plane Block and Serratus Anterior Plane Block for Breast Surgery: A Prospective Randomized Study
Brief Title: Ultrasound-guided Pectoral Nerve Blocks, Thoracic Erector Spinae Plane Block and Serratus Anterior Plane Block for Breast Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Salah El-Din Taha, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Management Department, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD276/9/24
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Ultrasound; Pectoral Nerve Blocks; Thoracic Erector Spinae Plane Block; Serratus Anterior Plane Block; Breast Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pectoral nerve block (PECS) (Experimental): Patients will receive pectoral nerve block (PECS).
  Interventions: Drug: Pectoral nerve block (PECS)
- Erector spinae plane block (ESP) (Experimental): Patients will receive erector spinae plane block (ESP).
  Interventions: Drug: Erector spinae plane block (ESP)
- Serratus anterior plane block (SAP) (Experimental): Patients will receive serratus anterior plane block (SAP).
  Interventions: Drug: Serratus anterior plane block (SAP)

INTERVENTIONS:
Drug: Pectoral nerve block (PECS) — Patients will receive pectoral nerve block (PECS).
  Other Names: Bupivacaine 0.25
  Arms: Pectoral nerve block (PECS)
Drug: Erector spinae plane block (ESP) — Patients will receive erector spinae plane block (ESP).
  Other Names: Bupivacaine 0.25
  Arms: Erector spinae plane block (ESP)
Drug: Serratus anterior plane block (SAP) — Patients will receive serratus anterior plane block (SAP).
  Other Names: Bupivacaine 0.25
  Arms: Serratus anterior plane block (SAP)

SUMMARY:
The study will compare ultrasound-guided Pectoral nerve block, Erector Spinae Plane block, and Serratus anterior plane block for pain management following elective breast surgeries

DETAILED DESCRIPTION:
Adequate acute postoperative pain control is important for patients undergoing breast surgery because the pain may be severe and longlasting. Surgical incision at the breast and axillary areas is associated with significant pain, with high incidence of acute pain progressing to chronic pain in 25% to 60% of patients. Post-mastectomy pain managed with opioids often lead to side effects of nausea and vomiting.

Regional anesthetic techniques are used in the current management of pain associated with breast surgeries .They attenuate surgical stress response , intraoperative consumption of opioid, prevent central sensitization and diminish postoperative pain.

The efficacy of fascial plane blocks like pectoral nerve block (PECS), serratus anterior plane block (SAP), and erector spinae plane block (ESP) has been proven in previous studies. These blocks require deposition of local anesthetic in an inter-fascial plane through which peripheral nerves travel.

The Pectoral nerve block relies upon the deposition the local anesthetic at the inter-fascial planes among the pectoralis major, minor, and serratus anterior muscles: it blocks the pectoral, the intercostobrachial, the intercostals III and VI, and the long thoracic nerves.

Erector Spinae Plane block is another interfacial plane block. It involves deposition of local anesthetic between erector spinae muscle and transverse process of T5 vertebrae and targets both dorsal and ventral rami of thoracic spinal nerves.

Serratus anterior plane block involves the injection of local anesthetic in 1 of the 2 fascial planes, superficial and deep to serratus anterior muscle at the level of the fifth rib in midaxillary line. The SAP block targets the lateral cutaneous branches of the thoracic intercostal nerves. The deep SAP block was found to have similar analgesic efficacy and technically easier and safer to perform as compared to the superficial SAP block.

ELIGIBILITY:
Inclusion Criteria:

• Age from 21 to 65 years old female, American Society of Anesthesiologists (ASA) physical status I or II, who will undergo breast surgeries under general anesthesia.

Exclusion Criteria:

* Patient refusal to participate in research.
* Body Mass Index (BMI) ≥35 kg/m2.
* Sensitivity to the intervention drugs.
* Coagulation abnormalities.
* Psychiatric disorder and communication difficulties.
* Chronic neurological disease.
* Any skin infection at the needle puncture site.
* Chest wall deformity

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the visual analogue scale (VAS) ≥ 4 to be repeated after 30 min if pain persists until the VAS< 4.

SECONDARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to 1st request for the rescue of analgesia (time from the end of surgery till first dose of morphine administrated) will be recorded.
Intraoperative fentanyl consumption | Intraoperatively
  Intraoperative fentanyl consumption will be recorded.Additional fentanyl bolus dosages of 0.5 µg/kg IV will be administered if mean arterial blood pressure and heart rate elevated more than 20% of the baseline (after exclusion of other causes).
Pain degree | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analogue scale (VAS) (20), from 0 to 10 (0 represents "no pain" while 10 represents "the worst pain imaginable").Rescue analgesia of morphine will be given as 3 mg bolus if the VAS ≥ 4 to be repeated after 30 min if pain persists until the VAS< 4. VAS will be assessed at 30min, 2, 6,12 and 24 h postoperatively
Mean arterial blood pressure | Till the end of surgery (Up to 24hours)
  Intraoperative hemodynamic parameters: Mean arterial blood pressure (MAP) will be recorded at baseline, after performing of block, and every 15 min till the end of surgery.
Heart rate | Till the end of surgery (Up to 24hours)
  Intraoperative hemodynamic parameters: Heart rate (HR) will be recorded at baseline, after performing of block, and every 15 min till the end of surgery.
Patient satisfaction | 24 hours Postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Adverse effects | 24 hours Postoperatively
  bradycardia, hypotension, nausea, vomiting, respiratory depression, hematoma at the site of injection, local anesthetic toxicity will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.